CLINICAL TRIAL: NCT04716894
Title: Effect of Itraconazole on the Pharmacokinetics of a Single Oral Dose of BI 474121 in Healthy Male Subjects (an Open-label, Two-period Fixed Sequence Design Study)
Brief Title: A Study in Healthy Men to Test How Itraconazole Influences the Amount of BI 474121 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1411-0010; 2019-003630-16 (EudraCT Number)
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequence: BI 474121 alone (Reference) - Itraconazole + BI 474121 (Test) (Experimental): Period 1:
  Reference (R) treatment: Healthy subjects received a single dose of 0.5 milligram (Powder for oral solution, 0.5 milligram (mg)/milliliter (mL) formulation) BI 474121 on day 1 of period 1.
  Period 2:
  Test (T) treatment: Healthy subjects received a daily dose of 200 milligram (oral solution, 10 mg/mL) Itraconazole for 14 days (days -3 - 11 of period 2) and a single dose of 0.5 milligram (Powder for oral solution, 0.5 milligram mg/mL formulation) BI 474121 on day 1 of period 2.
  BI 474121 administrations in treatment R and treatment T were separated by a wash-out period of at least 10 days.
  Administration of trial medication with 240 mL of water was performed after subjects had fasted overnight; fasting was to start no later than 10 hours before the scheduled dosing of BI 474121 or 9 hours before itraconazole administration.
  Interventions: Drug: BI 474121; Drug: Itraconazole

INTERVENTIONS:
Drug: BI 474121 — BI 474121 oral solution
Drug: Itraconazole — Itraconazole oral solution

SUMMARY:
The main objective of this trial is to investigate the effect on the exposure of BI 474121 in plasma when given as oral single dose together with multiple oral doses of itraconazole (Test, T) as compared to when given alone as oral single dose (Reference, R).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including blood pressure, pulse rate or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was an open-label, two-treatment, two-period, fixed-sequence design trial in healthy male subjects that explored the effect of multiple doses of itraconazole on the single-dose pharmacokinetics of BI 474121.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Sequence: BI 474121 Alone (Reference) - Itraconazole + BI 474121 (Test): Period 1:
  Reference (R) treatment: Healthy subjects received a single dose of 0.5 milligram (Powder for oral solution, 0.5 milligram (mg)/milliliter (mL) formulation) BI 474121 on day 1 of period 1.
  Period 2:
  Test (T) treatment: Healthy subjects received a daily dose of 200 milligram (oral solution, 10 mg/mL) Itraconazole for 14 days (days -3 to 11 of period 2) and a single dose of 0.5 milligram (Powder for oral solution, 0.5 milligram mg/mL formulation) BI 474121 on day 1 of period 2.
  BI 474121 administrations in treatment R and treatment T were separated by a wash-out period of at least 10 days.
  Administration of trial medication with 240 mL of water was performed after subjects had fasted overnight; fasting was to start no later than 10 hours before the scheduled dosing of BI 474121 or 9 hours before itraconazole administration.
Period: Period 1: BI 474121 Alone (Reference)
Arm/Group | Sequence: BI 474121 Alone (Reference) - Itraconazole + BI 474121 (Test)
Started | 14
Completed | 14
Not Completed | 0
Period: Period 2: Itraconazole Alone
Arm/Group | Sequence: BI 474121 Alone (Reference) - Itraconazole + BI 474121 (Test)
Started | 14
Treated | 13
Completed (Completed planned treatment) | 12
Not Completed | 2
Not completed — Not treated: positive alcohol test | 1
Not completed — COVID-19 related reason | 1
Period: Period 2: Itraconazole+BI 474121 (Test)
Arm/Group | Sequence: BI 474121 Alone (Reference) - Itraconazole + BI 474121 (Test)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were treated with at least one dose of study drug.
Arm/Group | Sequence: BI 474121 Alone (Reference) - Itraconazole + BI 474121 (Test)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 474121 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 474121 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞). Model used was an analysis of variance (ANOVA) model on the logarithmic scale. Data were log-transformed (natural logarithm) prior to fitting the ANOVA model. The effect 'subjects' was considered as random effect, whereas 'treatment' was considered as fixed effect.
Time Frame: Within 3 hours before and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 7, 8, 10, 12, 24, 34, 46, 70, 94, 118, 142 hours after BI 474121 administration in each period. In addition at 166, 190, 214, 238, 262 hours after BI 474121 administration in period 2.
Population: Pharmacokinetic parameter analysis set (PKS): all subjects who were treated with at least one dose of study drug and who provided at least one Pharmacokinetic (PK) endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
  Only subjects with non-missing values were included in the analyses.
Measure: Geometric Mean (Standard Deviation); unit: hours*nanomole/Liter
Groups:
- Reference (R) Treatment: BI 474121 Alone: Period 1: Reference (R) treatment: Healthy subjects received a single dose of 0.5 milligram (Powder for oral solution, 0.5 milligram (mg)/milliliter (mL) formulation) BI 474121 on day 1 of period 1.
  Administration of trial medication with 240 mL of water was performed after subjects had fasted overnight; fasting was to start no later than 10 hours before the scheduled dosing of BI 474121 administration.
- Test (T) Treatment: Itraconazole + BI 474121: Period 2: Test (T) treatment: Healthy subjects received a daily dose of 200 milligram (oral solution, 10 mg/mL) Itraconazole for 14 days (days -3 to 11 of period 2) and a single dose of 0.5 milligram (Powder for oral solution, 0.5 milligram mg/mL formulation) BI 474121 on day 1 of period 2.
  Administration of trial medication with 240 mL of water was performed after subjects had fasted overnight; fasting was to start no later than 10 hours before the scheduled dosing of BI 474121 or 9 hours before itraconazole administration.
Arm/Group | Reference (R) Treatment: BI 474121 Alone | Test (T) Treatment: Itraconazole + BI 474121
Number analyzed (Participants) | 13 | 12
hours*nanomole/Liter | NA (NA) — Adjusted Geometric Means = 67.09 Adjusted geometric standard error (gSE) = 1.07 | NA (NA) — Adjusted Geometric Means = 132.69 Adjusted geometric standard error (gSE) = 1.07
Statistical Analysis 1: Comparison: Reference (R) Treatment: BI 474121 Alone vs Test (T) Treatment: Itraconazole + BI 474121; Relative bioavailability. Model used was an analysis of variance (ANOVA) model on the logarithmic scale. Data were log-transformed (natural logarithm) prior to fitting the ANOVA model. The effect 'subjects' was considered as random effect, whereas 'treatment' was considered as fixed effect; Test type: Other; adjusted geometric mean (gMean) ratio(%) = 197.77, 90% CI 2-sided [187.90 to 208.15] — Ratio (%) = T/R*100. Intra-individual geometric coefficient of variation (gCV) = 7.0

2. Primary Outcome: Maximum Measured Concentration of BI 474121 in Plasma (Cmax)
Description: Maximum measured concentration of BI 474121 in plasma (Cmax). Model used was an analysis of variance (ANOVA) model on the logarithmic scale. Data were log-transformed (natural logarithm) prior to fitting the ANOVA model. The effect 'subjects' was considered as random effect, whereas 'treatment' was considered as fixed effect.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Nanomole/Liter
Arm/Group | Reference (R) Treatment: BI 474121 Alone | Test (T) Treatment: Itraconazole + BI 474121
Number analyzed (Participants) | 13 | 12
Nanomole/Liter | NA (NA) — Adjusted Geometric Means = 8.31 Adjusted geometric standard error (gSE) = 1.06 | NA (NA) — Adjusted Geometric Means = 11.92 Adjusted geometric standard error (gSE) = 1.07
Statistical Analysis 1: Comparison: Reference (R) Treatment: BI 474121 Alone vs Test (T) Treatment: Itraconazole + BI 474121; [analysis description as in outcome 1, analysis 1]; Test type: Other; adjusted geometric mean (gMean) ratio(%) = 143.38, 90% CI 2-sided [121.92 to 168.60] — Ratio (%) = T/R*100. Intra-individual geometric coefficient of variation (gCV) = 22.1

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 474121 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 474121 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz). Model used was an analysis of variance (ANOVA) model on the logarithmic scale. Data were log-transformed (natural logarithm) prior to fitting the ANOVA model. The effect 'subjects' was considered as random effect, whereas 'treatment' was considered as fixed effect.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Hours*nanomole/Liter
Arm/Group | Reference (R) Treatment: BI 474121 Alone | Test (T) Treatment: Itraconazole + BI 474121
Number analyzed (Participants) | 13 | 12
Hours*nanomole/Liter | NA (NA) — Adjusted Geometric Means = 64.53 Adjusted geometric standard error (gSE) = 1.07 | NA (NA) — Adjusted Geometric Means = 130.13 Adjusted geometric standard error (gSE) = 1.07
Statistical Analysis 1: Comparison: Reference (R) Treatment: BI 474121 Alone vs Test (T) Treatment: Itraconazole + BI 474121; [analysis description as in outcome 1, analysis 1]; Test type: Other; adjusted geometric mean (gMean) ratio(%) = 201.64, 90% CI 2-sided [192.23 to 211.52] — Ratio (%) = T/R*100. Intra-individual geometric coefficient of variation (gCV) = 6.5

ADVERSE EVENTS:
Time Frame: R treatment: first administration of BI 474121 until 7 days thereafter. Up to 7 days. T treatment: Itraconazole alone: first administration of itraconazole until time of BI 474121 administration OR until 3 days after last dose of itraconazole. Up to 6 days. T treatment: Itraconazole + BI 474121: BI 474121 administration in treatment period 2 until 3 days after the last administration of itraconazole OR 7 days after the BI 474121 administration in period 2, whatever is later. Up to 14 days.
Description: Treated set (TS): The treated set included all subjects who were treated with at least one dose of study drug.
Groups:
- Test (T) Treatment: Itraconazole Alone: Period 2: Test (T) treatment: Healthy subjects received a daily dose of 200 milligram (oral solution, 10 mg/mL) Itraconazole for 3 days (day -3 to day -1 of period 2).
  Administration of trial medication with 240 mL of water was performed after subjects had fasted overnight; fasting was to start no later than 9 hours before itraconazole administration.
- Test (T) Treatment: Itraconazole + BI 474121: Period 2: Test (T) treatment: Healthy subjects received a daily dose of 200 milligram (oral solution, 10 mg/mL) Itraconazole and a single dose of 0.5 milligram (Powder for oral solution, 0.5 milligram mg/mL formulation) BI 474121 on day 1 of period 2. This arm only considers the time when Itraconazole was given together with BI 474121 during period 2 (day 1 to 11 of period 2).
  Administration of trial medication with 240 mL of water was performed after subjects had fasted overnight; fasting was to start no later than 10 hours before the scheduled dosing of BI 474121 or 9 hours before itraconazole administration.
Arm/Group | Reference (R) Treatment: BI 474121 Alone | Test (T) Treatment: Itraconazole Alone | Test (T) Treatment: Itraconazole + BI 474121
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 2/14 | 0/13 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reference (R) Treatment: BI 474121 Alone (N=14) | Test (T) Treatment: Itraconazole Alone (N=13) | Test (T) Treatment: Itraconazole + BI 474121 (N=12)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT04716894/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT04716894/SAP_001.pdf